CLINICAL TRIAL: NCT00633256
Title: The Effect of Cycloserine on Smoking Behavior in Nicotine Dependent Smokers.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: VA Connecticut Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, James Poling, Research Scientist, Yale University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 0601001031
Record Dates: First submitted 2008-02-29; First posted 2008-03-11 (Estimated); Results first posted 2012-04-11 (Estimated); Last update posted 2012-04-11 (Estimated); Status verified 2012-03

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking | interventions — Cycloserine; Tacrine; Isoniazid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cycloserine (Experimental): 50 mg cycloserine
  Interventions: Drug: Cycloserine
- Placebo (Sham Comparator): Matched placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cycloserine — 50 mg Cycloserine given in two separate experimental sessions separated by approximately one week.
  Other Names: Closina Aspen, Austral.; Cycloserine Capsules USP 29; Cycloserine (TM)King, UK; D-cycloserin IFET (IFET), Gr.; Proserine Hawon, Thai.; Seromycin - 250 MG - Capsule Dura Pharmaceuticals; Seromycin - 250 MG - Oral Capsule Eli Lilly; Seromycin (FM) Lilly, Canad.; Seromycin Dura, USA; Seromycin Lilly, Hong Kong; Seromycin With Isoniazid - 250 MG - Capsule Eli Lilly; Siklocap
  Arms: Cycloserine
Drug: Placebo — Matched placebo for subjects randomized to placebo arm. Given in two experimental sessions separated by approximately one week.
  Arms: Placebo

SUMMARY:
A total of 20 subjects will participate in this four week, between groups, double-blind, placebo controlled study. Subjects will participate in two experimental sessions separated by approximately one week. Subjects will be randomized to receive either 50 mg cycloserine or placebo combined with cue exposure. Several physiological and subjective outcome measures (e.g., heart rate, blood pressure, galvanic skin response) will be obtained during the sessions. Experimental sessions will last approximately 4.5 hours with follow-up sessions lasting approximately thirty minutes. Our aims are:

1. To examine the effect of cycloserine vs. placebo on extinction of smoking cue reactivity in overnight abstinent smokers. Reactivity to smoking cues will be captured with self-report smoking urges and physiological measures (heart rate, blood pressure, and skin conductance).

   We hypothesize that cycloserine, relative to placebo, will facilitate extinction of smoking cue reactivity.
2. To examine the effect of cycloserine vs. placebo when combined with two 4.5 hour laboratory cue exposure training sessions, on smoking behavior in smokers. Smoking behavior will be measured with self-report smoking and saliva cotinine levels.
3. To examine the effect of cycloserine vs. placebo on memory performance in nicotine dependent smokers. Memory performance will be measured with verbal learning, recognition and recall tasks.

4) To examine the safety and tolerability of cycloserine treatment in smokers. We hypothesize that cycloserine will be well tolerated by smokers.

ELIGIBILITY:
Inclusion Criteria:

* female and male smokers, aged 18 to 55 years;
* history of smoking daily for the past 12 months, at least 10 cigarettes daily;
* CO level > 10ppm;
* for women: not pregnant as determined by pregnancy screening, nor breast feeding, and using acceptable birth control methods other than OCP;
* Non-treatment seeking nicotine dependent smokers.

Exclusion Criteria:

* history of heart disease, renal or hepatic diseases or other medical conditions that the physician investigator deems as contraindicated for the patient to be in the study;
* regular use of psychotropic medication (antidepressants, antipsychotics, or anxiolytics) and/or recent psychiatric diagnosis and treatment for Axis I disorders including major depression, bipolar affective disorder, schizophrenia and panic disorder within the past year;
* current dependence on alcohol or on drugs other than nicotine;
* regular use of any other tobacco products than cigarettes, including smokeless tobacco and nicotine products;
* allergy to cycloserine;
* subjects with epilepsy or a history of seizures;
* Treatment seeking nicotine dependent smokers.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2006-12; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Poling, Ph.D., Principal Investigator — Yale University
Locations (1):
- West Haven VA, West Haven, Connecticut, United States

REFERENCES:
- [Background] Santa Ana EJ, Rounsaville BJ, Frankforter TL, Nich C, Babuscio T, Poling J, Gonsai K, Hill KP, Carroll KM. D-Cycloserine attenuates reactivity to smoking cues in nicotine dependent smokers: a pilot investigation. Drug Alcohol Depend. 2009 Oct 1;104(3):220-7. doi: 10.1016/j.drugalcdep.2009.04.023. Epub 2009 Jul 9. PMID 19592176

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cycloserine | Placebo
Started | 12 | 13
Completed | 8 | 10
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cycloserine | Placebo | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 13 | 25
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 41.1 (6.2) | 41.5 (11.5) | 41.3 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 6 | 6 | 12
Region of Enrollment [Number; unit: participants]
  United States | 12 | 13 | 25

OUTCOME MEASURES:

1. Primary Outcome: Cigarettes Smoked Per Day
Description: The number of cigarettes smoked per day at the 1 week follow up time point.
Time Frame: 1 week follow-up
Population: The number of participants used for analysis were those who completed the 4-week follow-up timepoint.
Measure: Mean (Standard Deviation); unit: Cigarettes per day
Arm/Group | Cycloserine | Placebo
Number analyzed (Participants) | 8 | 8
Cigarettes per day | 10.3 (6.3) | 13.9 (12.7)

2. Secondary Outcome: Cigarettes Smoked Per Day
Description: The number of cigarettes smoked per day at the 4-week follow up timepoint.
Time Frame: 4 Week Followup
Population: The number of subjects in the study at the 4-week timepoint.
Measure: Mean (Standard Deviation); unit: Cigarettes per day
Arm/Group | Cycloserine | Placebo
Number analyzed (Participants) | 8 | 8
Cigarettes per day | 9.9 (7.7) | 11.0 (9.2)

3. Secondary Outcome: Urinary Cotinine Level
Description: Urinary Cotinine level at the 4-week follow up timepoint
Time Frame: 4 Week Follow-up Timepoint
Population: Subjects used for analysis are those who reached the 4 week followup timepoint.
Measure: Mean (Standard Deviation); unit: Mean ng/ml
Arm/Group | Cycloserine | Placebo
Number analyzed (Participants) | 8 | 8
Mean ng/ml | 1645.5 (1180.8) | 2062.6 (1091.1)

ADVERSE EVENTS:
Arm/Group | Cycloserine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 0/12 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes